CLINICAL TRIAL: NCT03070106
Title: Assessment of Diabetes Control, Cost of Care, and Quality of Life Utilizing a Functional Medicine Approach in Addition to Usual Care Vs. Usual Care Alone
Brief Title: Diabetes: Functional Medicine Approach Vs. Usual Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keren Zhou (Other)
Responsible Party: Sponsor-Investigator, Keren Zhou, Associate Staff, Endocrinology and Metabolism Institute, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1339
Record Dates: First submitted 2017-02-20; First posted 2017-03-03 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Diabetes; Type 2 Diabetes; Type 2 Diabetes Treated with Insulin
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Comparison between the functional medicine (FM) group and the usual care group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): usual care delivered by an endocrinologist
- Functional Medicine + Usual Care (Active Comparator): Functional Medicine in addition to usual care delivered by an endocrinologist
  Interventions: Dietary Supplement: Functional Medicine

INTERVENTIONS:
Dietary Supplement: Functional Medicine — Subjects randomized to the Functional Medicine plus the usual care arm will receive nutrition therapy and dietary supplements. Functional Medicine labs will be used in part to determine which supplements will be prescribed.
  Arms: Functional Medicine + Usual Care

SUMMARY:
A Functional Medicine (FM) approach to diabetes care focuses on identifying and treating the etiologies for "imbalances in the core physiological systems."(1) If underlying triggers and imbalances can be identified, the FM approach to addressing "root causes"(1) can be utilized through the use of specialized testing to treat and potentially reverse diabetes. If the FM approach is successful, the impact on diabetes disease burden as well as diabetes-associated health care costs could be significant. This project will assess the clinical as well as cost effectiveness of a FM approach to diabetes care compared to a usual care approach for patients with diabetes on insulin for 5 years or less.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, open-label clinical trial with a 1:1 randomization of patients with diabetes who have been on insulin less than 5 years to receive either Functional Medicine care in addition to usual care or to continue usual care delivered by an endocrinologist. The total number of patients planned for enrollment is 90, 45 in each arm. Patient recruitment will begin in the Cleveland Clinic main campus Endocrinology clinics and may later include Endocrinology practices at other Cleveland Clinic Health System sites.

Following voluntary informed consent, study subjects will complete a screening/baseline visit. After this visit, patients will be randomized to continuing usual care delivered by endocrinologists or to FM plus usual care. Once randomization occurs, the patient will continue to remain under the care of their endocrinologist and any other usual physicians. If randomized to the FM plus usual care group, subjects will receive additional care through a functional medicine physician.

A stratified randomization procedure will be used to allocate patients into the two groups according to the strata: Total Daily Insulin dose < = 50 units vs. > 50 units.

All subjects: In addition to usual care provided by the endocrinologist, study visits will occur at screening/baseline, 6 months, 12 months and 24 months. Lab data/Biometrics (if not recorded within 1 month time frame) will be obtained at this time. Quality of life instruments (Diabetes Distress Scale, SPADE, PHQ-9 and MSQ; Appendices D, E, F and G) will also be administered. At baseline, the 12 month visit, and the 24 month visit, a Body Fat Analysis by Bioelectrical impedance analysis (BIA) will be performed. There will also be 10 cc of blood collected for plasma and serum samples as well as 10 cc of urine and approximately 1 gram of stool for the bio repository if patient agrees to provide the samples.

Usual care subjects only: Subjects randomized to the usual care arm will receive a nutritional education session.

FM plus usual care subjects only: Subjects randomized to the FM plus usual care arm will be evaluated using the functional medicine approach to diabetes outlined in the Functional Medicine Diagnostic and Treatment Approach to Type 2 Diabetes Mellitus and Cardio-Metabolic Syndrome. Subjects randomized to the FM plus usual care arm will also receive nutrition therapy and dietary supplements. These will be prescribed and monitored at all Functional Medicine study visits. An estimated total of 50ml of blood will be collected from those subjects in this arm of the study at each designated visit. In addition, subjects may be asked to provide a urine and stool sample. Functional Medicine labs will be used in part to determine which supplements will be recommended.

ELIGIBILITY:
Inclusion Criteria:

* Seen in the Cleveland Clinic Main Campus Endocrinology Clinics
* Diagnosis of Type 2 Diabetes
* Insulin treatment for at least 12 months, but for less than 96 months
* Total Daily Insulin Dose <= 150 units

Exclusion Criteria:

* Positive glutamate decarboxylase antibody
* C peptide < 0.8 ng/ml
* Use of Insulin Pump for diabetes treatment
* HbA1c > 12%
* History of Diabetic Ketoacidosis (DKA) defined by patient report or any emergency department visits or hospitalization for DKA
* Pregnancy
* Breastfeeding
* Known diagnosis of Cognitive Impairment or Dementia
* Estimated Glomerular Filtration Rate < 45 ml/min/1.73m
* Congestive Heart Failure New York Heart Association (NYHA) Functional Class III or IV
* Active Malignancy
* Human Immunodeficiency Virus infection on treatment with medications
* Treatment with steroids (medication related diabetes)
* Treatment with antipsychotics (medication related diabetes)
* Abnormal baseline Complete Blood Count
* Liver Function tests > 3 times upper limit of normal, Viral Hepatitis, or Elevated Liver Function tests of Unclear Etiology
* Currently participating in a supervised diet program through Department of Endocrinology
* Currently participating in any other research study, such as 15-1134: Prospective Validation of Predictive Tool study through Department of Endocrinology
* Treatment with Coumadin (warfarin)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-03-05 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects in each study arm discontinuing insulin use with no increase in Hemoglobin A1c | Baseline to 6 months
  Discontinuation of insulin-no increase in Hemoglobin A1c-6 months
Number of subjects in each study arm discontinuing insulin use with no increase in Hemoglobin A1c | Baseline to 12 months
  Discontinuation of insulin-no increase in Hemoglobin A1c-12 months
Number of subjects in each study arm discontinuing insulin use with Hemoglobin A1c <7% | Baseline to 6 months
  Discontinuation of insulin-Hemoglobin A1c <7%-6 months
Number of subjects in each study arm discontinuing insulin use with Hemoglobin A1c <7% | Baseline to 12 months
  Discontinuation of insulin-Hemoglobin A1c <7%-12 months

SECONDARY OUTCOMES:
Number of subjects in each study arm reducing insulin use (units) with no increase in Hemoglobin A1c | Baseline to 6 months
  Reduction in insulin use-no increase in Hemoglobin A1c-6 months
Number of subjects in each study arm reducing insulin use (units) with no increase in Hemoglobin A1c | Baseline to 12 months
  Reduction in insulin use-no increase in Hemoglobin A1c-12 months
Number of subjects in each study arm reducing insulin use (units) with Hemoglobin A1c <7% | Baseline to 6 months
  Reduction in insulin use-Hemoglobin A1c <7%-6 months
Number of subjects in each study arm reducing insulin use (units) with Hemoglobin A1c <7% | Baseline to 12 months
  Reduction in insulin use-Hemoglobin A1c <7%-12 months
Reduction in the number of units of insulin used by subjects in each study arm with no increase in Hemoglobin A1c | Baseline to 6 months
  Reduction in number of insulin units-no increase in Hemoglobin A1c-6 months
Reduction in the number of units of insulin used by subjects in each study arm with no increase in Hemoglobin A1c | Baseline to 12 months
  Reduction in number of insulin units-no increase in Hemoglobin A1c-12 months
Reduction in the number of units of insulin used by subjects in each study arm with Hemoglobin A1c <7% | Baseline to 6 months
  Reduction in number of insulin units-Hemoglobin A1c <7%-6 months
Reduction in the number of units of insulin used by subjects in each study arm with Hemoglobin A1c <7% | Baseline to 12 months
  Reduction in number of insulin units-Hemoglobin A1c <7%-12 months
Total reduction in Hemoglobin A1c percentage for subjects in each study arm | Baseline to 6 months
  Evaluate diabetes control using subject hemoglobin A1c values-6 months
Total reduction in Hemoglobin A1c percentage for subjects in each study arm | Baseline to 12 months
  Evaluate diabetes control using subject hemoglobin A1c values-12 months
Change in low density lipoprotein [LDL] (mg/dL) for subjects in each study arm | Baseline to 6 months
  Evaluate cardiovascular risk factor using Low density lipoprotein values-6 months
Change in low density lipoprotein [LDL] (mg/dL) for subjects in each study arm | Baseline to 12 months
  Evaluate cardiovascular risk factor using Low density lipoprotein values-12 months
Change in high density lipoprotein [HDL] (mg/dL) for subjects in each study arm | Baseline to 6 months
  Evaluate cardiovascular risk factor using High density lipoprotein (HDL)-6 months
Change in high density lipoprotein [HDL] (mg/dL) for subjects in each study arm | Baseline to 12 months
  Evaluate cardiovascular risk factor using High density lipoprotein (HDL)-12 months
Change in systolic blood pressure (mm/Hg) for subjects in each study arm | Baseline to 6 months
  Evaluate cardiovascular risk factor using systolic blood pressure-6 months
Change in systolic blood pressure (mm/Hg) for subjects in each study arm | Baseline to 12 months
  Evaluate cardiovascular risk factor using systolic blood pressure-6 months
Change in body weight (kg) for subjects in each study arm | Baseline to 6 months
  Evaluate cardiovascular risk factor using Body weight-6 months
Change in body weight (kg) for subjects in each study arm | Baseline to 12 months
  Evaluate cardiovascular risk factor using Body weight-12 months
Number of hypoglycemic episodes occurring in subjects in each study arm | Baseline to 6 months
  Evaluate the frequency of hypoglycemia-6 months
Number of hypoglycemic episodes occurring in subjects in each study arm | Baseline to 12 months
  Evaluate the frequency of hypoglycemia-12 months
Cost (dollars) of health care for subjects in each study arm | Baseline to 12 months
  Cost of office visits, emergency room visits, hospital admissions, medication costs
Reduction in the total number of medications required for subjects in each study arm | Baseline to 12 months
  Reduction in medication requirements
Change in the subject's overall score on the Diabetes Distress Scale in each study arm | Baseline to 6 months
  Evaluate quality of life ratings using the Diabetes Distress Scale-6 months
Change in the subject's overall score on the Diabetes Distress Scale in each study arm | Baseline to 12 months
  Evaluate quality of life ratings using the Diabetes Distress Scale-12 months
Change in the subject's T-Score on the SPADE survey in each study arm | Baseline to 6 months
  Evaluate quality of life ratings using the general quality of life instrument (SPADE)-6 months
Change in the subject's T-Score on the SPADE survey in each study arm | Baseline to 12 months
  Evaluate quality of life ratings using the general quality of life instrument (SPADE)-12 months
Change in the subject's score on the Medical Symptom Questionnaire (MSQ) in each study arm | Baseline to 6 months
  Evaluate quality of life ratings using the Medical Symptom Questionnaire (MSQ)-6 months
Change in the subject's score on the Medical Symptom Questionnaire (MSQ) in each study arm | Baseline to 12 months
  Evaluate quality of life ratings using the Medical Symptom Questionnaire (MSQ)-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Betul Hatipoglu, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No